CLINICAL TRIAL: NCT00876720
Title: Effectiveness of Combined Frontal and Temporal Repetitive Transcranial Magnetic Stimulation (rTMS) in Patients With Chronic Tinnitus
Brief Title: Effectiveness Repetitive Transcranial Magnetic Stimulation (rTMS) in Patients With Chronic Tinnitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Regensburg (Other)
Responsible Party: Berthold Langguth, MD, University of Regensburg, Dept of Psychiatry
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Uni-Reg-rTMS-Tinnitus-01
Record Dates: First submitted 2009-04-06; First posted 2009-04-07 (Estimated); Last update posted 2010-11-15 (Estimated); Status verified 2010-11

CONDITIONS: Tinnitus
Keywords: Tinnitus; chronic subjective tinnitus; transcranial magnetic stimulation; sensation disorders; hearing disorders
MeSH Terms: conditions — Tinnitus; Sensation Disorders; Hearing Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Combined frontal and temporal transcranial magnetic stimulation
  Interventions: Device: rTMS - Intervention 1
- 2 (Experimental): Temporal transcranial magnetic stimulation
  Interventions: Device: rTMS - Intervention 2

INTERVENTIONS:
Device: rTMS - Intervention 1 — Experimental repetitive transcranial magnetic stimulation (Alpine Biomed Mag Pro Option): 2000 stimuli of 20Hz rTMS over the left DLPFC (110% motor threshold) followed by 2000 stimuli of 1 Hz rTMS over the left temporal cortex DLPFC (110% motor threshold)
  Arms: 1
Device: rTMS - Intervention 2 — Experimental repetitive transcranial magnetic stimulation (Alpine Biomed Mag Pro Option): 2000 stimuli of 1 Hz rTMS over the left temporal cortex DLPFC (110% motor threshold)
  Arms: 2

SUMMARY:
Transcranial Magnetic Stimulation is used to modulate the auditory neural pathways caused by hearing loss and leading to the phantom auditory perception of sound in the absence of an external or internal acoustic stimulus.

DETAILED DESCRIPTION:
Tinnitus is the phantom auditory perception of sound in the absence of an external or internal acoustic stimulus. It is a frequent problem which can interfere significantly with the ability to lead a normal life. Treatment is difficult. Most available therapies focus on habituation rather than treating the cause. Tinnitus is thought to be generated in the brain, as a result of functional reorganization of auditory neural pathways and tonotopic maps in the central auditory system, following damage to the peripheral auditory system. Low-frequency rTMS has been investigated for the treatment of hyperexcitability disorders such as auditory hallucinations and tinnitus. Pilot data indicate that the beneficial effect of low-frequency rTMS can be enhanced by high frequency rTMS of the left dorsolateral prefrontal cortex (DLPFC). In the proposed study we investigate whether high frequency rTMS of the DLPFC improves therapeutic efficacy of low-frequency rTMS on tinnitus in a controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of subjective chronic tinnitus
* Duration of tinnitus more than 3 months

Exclusion Criteria:

* Objective tinnitus
* Treatable cause of the tinnitus
* Involvement in other treatments for tinnitus at the same time
* Clinically relevant psychiatric comorbidity
* Clinically relevant unstable internal or neurological comorbidity
* History of or evidence of significant brain malformation or neoplasm, head injury
* Cerebral vascular events
* Neurodegenerative disorder affecting the brain or prior brain surgery;
* Metal objects in and around body that can not be removed
* Pregnancy
* Alcohol or drug abuse
* Prior treatment with TMS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2009-04; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
tinnitus severity as measured by the Tinnitus Questionnaire of Goebel and Hiller | Baseline, Day 12

CONTACTS AND LOCATIONS:
Overall Officials: Berthold Langguth, MD, Principal Investigator — University of Regensburg-Dept of Psychiatry
Locations (1):
- University of Regensburg - Dept of Psychiatry, Regensburg, Bavaria, Germany

REFERENCES:
- See also: Tinnitus Research and Treatment Center at the University of Regensburg — http://www.tinnituszentrum-regensburg.de/index.php